CLINICAL TRIAL: NCT02332226
Title: The PIFBO-study: Person-centred Information to Parents in Paediatric Oncology - A Randomized Controlled Trial Based Upon a Conceptual Framework for Patient Education
Brief Title: The PIFBO-study: Person-centred Information to Parents in Paediatric Oncology
Acronym: PIFBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University of Skövde (Other)
Responsible Party: Principal Investigator, Anders Ringnér, PhD, Senior lecturer, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PR2013-0086
Record Dates: First submitted 2014-12-11; First posted 2015-01-06 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Stress; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Representational approach (Experimental): Four sessions with a nurse. For each session, the parent identifies an area where he/she needs more information. The nurse and the parent jointly survey the parent's knowledge of the area and discusses consequences of knowledge gaps or misunderstandings. Then, new information is introduced and benefits from the new information is discussed.
  Interventions: Behavioral: Representational approach
- Control (No Intervention): Standard care as per ward protocol.

INTERVENTIONS:
Behavioral: Representational approach — Representational approach to patient education
  Arms: Representational approach

SUMMARY:
The aim of this project is to evaluate a person-centred informational intervention aimed at parents of children with cancer.

The following hypotheses will be tested: an informational intervention emanating from the parents' self-identified needs is associated to decreased illness-related parenting stress, decreased post-traumatic stress symptoms, increased received knowledge, decreased anxiety, decreased depression, increased satisfaction with information, and decreased number of health care contacts in parents.

DETAILED DESCRIPTION:
BACKGROUND

Parents of children with cancer have great information needs and report that these are not always met. Psychosocial suffering such as stress and anxiety is also common in this group.

INTERVENTION

The intervention in this study builds upon the representational approach for patient education. It emanates from Leventhal's theories about illness representation and educational theories about conceptual change. Central elements in the approach are parental choice of information topics of interest, and a thorough assessment of present parental knowledge before information is given. Each parent in the intervention arm gets four sessions with an intervention nurse.

DESIGN AND METHODS

The study comprises a multi-centre randomized controlled trial with two parallel arms with a 1:1 allocation ratio. One arm will receive the intervention and the other standard care according to local routines at each ward. The effect will be measured with validated instrument which are answered on a web platform. Complementary to the quantitative evaluation, we will perform a process evaluation aiming at understanding the change mechanisms, treatment fidelity, dose delivered, contextual factors of importance and how the intervention further could be optimized.

ELIGIBILITY:
Inclusion Criteria:

Being a parent of a child that

1. is diagnosed with a first time occurrence of a malignancy that is curatively treated and
2. was diagnosed two months ago.

   Further parents must be
3. able to talk, read and write Swedish enough to be able to participate without an interpreter.

Exclusion Criteria:

* None specific.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2019-07 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Pediatric Inventory for Parents (compare the mean scoring) | baseline up to one year post intervention
  An instrument with 42 items measuring both frequency and intensity of stressors related to having a chronically ill child.

SECONDARY OUTCOMES:
Impact of Event Scale-Revised (compare the mean scoring) | baseline up to one year post intervention
  22 items measuring posttraumatic stress symptoms.
Kowledge expectations of significant others and Received knowledge of significant others (compare the mean scorings) | baseline up to one year post intervention
  Two instruments measuring 40 areas of knowledge with respect to expectations and fulfilment.
Anxiety and depression (compare the mean scoring) | baseline up to one year post intervention
  Seven-point visual-digital scales.
Satisfaction with information (compare the mean scoring) | baseline up to one year post intervention
  Seven-point visual-digital scales.
Number of health care contacts | baseline up to one year post intervention
Experiences with your Health Care Provider (compare the mean scoring) | baseline up to one year post intervention
  15 items measuring the caring relationship with a health care provider

CONTACTS AND LOCATIONS:
Overall Officials: Anders Ringnér, PhD, Principal Investigator — Umeå University
Locations (2):
- Sweden (2):
  - Skåne University Hospital, Lund
  - Umeå University Hospital, Umeå

REFERENCES:
- [Background] Ringner A, Karlsson S, Hallgren Graneheim U. A person-centred intervention for providing information to parents of children with cancer. Experiences and effects. Eur J Oncol Nurs. 2015 Jun;19(3):318-24. doi: 10.1016/j.ejon.2014.10.012. Epub 2014 Nov 4. PMID 25466827
- [Derived] Ringner A, Bjork M, Olsson C. What Was on the Parents' Minds? Changes Over Time in Topics of Person-Centred Information for Mothers and Fathers of Children with Cancer. Compr Child Adolesc Nurs. 2023 Jun;46(2):114-125. doi: 10.1080/24694193.2023.2168790. Epub 2023 Feb 22. PMID 36811905
- [Derived] Ringner A, Bjork M, Olsson C. Effects of Person-Centered Information for Parents of Children With Cancer (the PIFBO Study): A Randomized Controlled Trial. J Pediatr Hematol Oncol Nurs. 2023 Nov-Dec;40(6):400-410. doi: 10.1177/27527530221115860. Epub 2023 Feb 2. PMID 36731493
- [Derived] Ringner A, Bjork M, Olsson C, Graneheim UH. Person-centred information to parents in paediatric oncology (the PIFBO study): A study protocol of an ongoing RCT. BMC Nurs. 2015 Dec 21;14:69. doi: 10.1186/s12912-015-0120-8. eCollection 2015. PMID 26770070